CLINICAL TRIAL: NCT00983528
Title: A Phase I/II Study of Alemtuzumab and Clofarabine for Relapsed or Refractory Acute Lymphoblastic Leukemia
Brief Title: Alemtuzumab and Clofarabine for Relapsed or Refractory Acute Lymphoblastic Leukemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Support withdrawn due to slow accrual
Sponsor: University of California, San Diego (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090331
Record Dates: First submitted 2009-09-23; First posted 2009-09-24 (Estimated); Results first posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-07

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: cancer; lymphoblastic; leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasms; Leukemia | interventions — Alemtuzumab; Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Alemtuzumab — 3mg day 1,10mg day 2, 30mg day 3, 30mg day 5, 30mg day 8, then three times per calendar week thereafter for a total 12- 30mg doses
  Other Names: Campath
Drug: Clofarabine — Dose Escalation
  Cycle 1 (30 days or until alemtuzumab completed) Clofarabine 10,20,30 or 40 mg/m2 days 5-9
  Cycle 2 and subsequent cycles (administered no more frequently than every 28 days) 10,20,30 or 40 mg/m2 days 1-5
  Other Names: Clolar

SUMMARY:
Clofarabine is approved by the FDA for the treatment of pediatric patients (1 to 21 years of age) with relapsed or refractory ALL. Alemtuzumab is approved by the FDA for treatment of B-cell chronic lymphocytic leukemia (B-CLL) in patients over the age of 18. These drugs have been used to treat patients with leukemia in other research studies like this one. Both drugs have individually been administered to adult patients with ALL with acceptable toxicity profiles. This study will evaluate the combination of clofarabine and alemtuzumab when administered to adult patients with relapsed or refractory ALL. Primary objectives of the study is to determine the maximum tolerated dose of clofarabine when administered with alemtuzumab, evaluate the safety of the combination, and assess for activity of the combination by evaluating response rate, effect on ALL progenitor cell population, and patients who are able to bridge to transplant.

DETAILED DESCRIPTION:
The strategy for treating relapsed and refractory adult ALL patients is through reinduction chemotherapy followed by allogeneic stem cell transplantation, provided that the toxicity of the salvage regimen is acceptable. However, this leukemia is characterized as being highly refractory to standard chemotherapy and therefore novel therapeutic approaches are desperately needed. Clofarabine is a second generation nucleoside analog FDA approved for the treatment of relapsed and refractory pediatric ALL. Clofarabine has been administered to adult patients with hematologic malignancies with an acceptable toxicity profile with 8% of relapsed ALL patients attaining a complete response (CR). The maximum tolerated dose (MTD) of clofarabine IV in adult patients has been determined to be 40 mg/m2/day for 5 consecutive days, which is lower than the tolerable daily dose for pediatric patients, 52 mg/m2/day. More recently, Karp and colleagues reported their experience with clofarabine in combination with cyclophosphamide in 18 patients with refractory acute leukemias. Encouraging responses were seen in the refractory ALL patients with 67% (4/6) patients experiencing a CR. Toxicity did not allow dose escalation of clofarabine and the MTD was defined as 10 mg/m2 administered over 6 non-consecutive days when combined with cyclophosphamide 200-400mg/m2 over a total of 7 days per cycle. As such, we are conservatively evaluating a clofarabine dose of 20mg/m2 for five days with a dose de-escalation step if there is dose limiting toxicity.

The addition of monoclonal antibody therapy is an attractive approach in the treatment of relapsed and refractory ALL since it targets both B and T progenitor ALL subtypes and has different mechanisms of action and side effects than chemotherapy. Alemtuzumab is a humanized monoclonal antibody to CD52 which is expressed on the majority of neoplastic lymphocytes, including 70% of ALL and 100% of Philadelphia positive ALL. The CALGB evaluated alemtuzumab as consolidation in front-line therapy for patients with ALL and demonstrated feasibility and found alemtuzumab administration at 30mg subcutaneously administered for 12 doses to be safe and well tolerated in a frontline consolidation setting in ALL. In the present protocol targeting refractory and relapsed ALL patients, the maximal alemtuzumab dose will be 30 mg as in Stock's study, but will be administered intravenously in order to improve the induction chemotherapy pharmacokinetics. Premedication with dexamethasone, benadryl, and acetaminophen will be given to all patients prior to alemtuzumab infusion to prevent infusional reactions associated with intravenous dosing.

The combination of purine analogs and alemtuzumab have been administered simultaneously safely with promising additive activity in other relapsed and refractory lymphocytic leukemias. A recent case series reported patients with relapsed and/or refractory ALL who failed several induction chemotherapies to achieve complete responses to fludarabine and alemtuzumab combination regimens. All patients were able to proceed to allogeneic SCT with refractory ALL patient relapsing at 8 months while relapsed patients remain in remission at 6 and 24 months.

Other approaches utilizing combination chemotherapy have failed to demonstrate consistent activity that would qualify them as standard of care. Therefore the standard of care for patients with relapsed and refractory ALL is enrollment into clinical trials.

All patients will receive alemtuzumab in a dose escalation fashion (3, 10, 30mg). Successive escalating doses will be administered if the previous dose is tolerated. Previously, Stock et al established the safety of 12 doses of 30mg of alemtuzumab in ALL. The treatment regimen is designed to have alemtuzumab administered prior to administration of clofarabine to allow dose escalation of the monoclonal antibody and decrease confounding acute toxicities such as infusion reactions and cytokine release. Clofarabine dose is modeled after previous trials in adult and pediatric ALL. The starting dose of clofarabine is lower than standard phase II doses for adult hematologic malignancy to conservatively evaluate tolerability and toxicity of clofarabine in combination with alemtuzumab. Alemtuzumab dosing will be limited to a total of 12. However, patients can continue with additional cycles of clofarabine if they do not show progressive disease or have unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed written informed consent. If a patient is under the 18 years of age the parent or the guardian will also need to provide written informed consent.
2. Diagnosis of ALL (B or T lineage) who have received therapy with at least 1 but not more than 3 prior different induction regimens and have been deemed to have relapse or refractory disease. The phase II component of the study enrollment will be limited to 2 different prior induction regimens if patients are older than 30 years.
3. ALL lymphoblasts with CD52 expression on at least 10% on lymphoblasts.
4. Age >= 16 years of age.
5. ECOG PS 0-2.
6. Have adequate renal and hepatic functions.
7. Subject or their patient or guardian is capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent.
8. Female patients of childbearing potential must have a negative serum pregnancy test within 2 weeks prior to enrollment.
9. Male and female patients must use an effective contraceptive method during the study and for a minimum of 6 months after study treatment. Subjects 16 and 17 years old must also adhere to effective contraception methods or abstinence during the study and for a minimum of 6 months after study and the nature of contraception or abstinence must be documented.
10. CMV PCR negative prior to enrollment

Exclusion Criteria:

1. Current concomitant chemotherapy, radiation therapy, or immunotherapy other than as specified in the protocol.
2. Use of investigational agents within 30 days or any anticancer therapy within 2 weeks before study entry with the exception of hydroxyurea, CNS treatment or prophylaxis, or tyrosine kinase inhibitors for individuals with Philadelphia chromosome positive ALL. The patient must have recovered from all acute toxicities from any previous therapy.
3. Lack of bone marrow or blood involvement by leukemia such as a documented CNS or testicular only relapse.
4. Have any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver, or other organ system that may place the patient at undue risk to undergo treatment.
5. Patients with any known or suspected Hepatitis B, C and HIV infections.
6. Patients with a systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
7. Pregnant or lactating patients.
8. Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - UCSD Medical Center, San Diego, California
  - Rady Children's Hospital, San Diego, California

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study enrolled six participants, but no participants completed study. Study was terminated due to slow accrual. All study data is reported by all participants since no data was analyzed due to study termination.
Groups:
- Alemtuzumab and Clofarabine: Alemtuzumab: Dose escalation (3mg, 10mg, to 30mg) Clofarabine: Maximum Tolerated Dose (10 mg/m2, 20 mg/m2, 30mg/m2, to 40 mg/m2 days 5-9)
Period: Overall Study
Arm/Group | Alemtuzumab and Clofarabine
Started | 6
Completed | 0
Not Completed | 6
Not completed — Death | 4
Not completed — Lost to Follow-up | 1
Not completed — Study Terminated | 1

BASELINE CHARACTERISTICS:
Population: Study enrolled six participants, but no participants completed study. Study was terminated due to slow accrual. All study data is reported by all participants since no data was analyzed due to study termination.
Arm/Group | Alemtuzumab and Clofarabine
Number analyzed (Participants) | 6
Age, Continuous [Mean (Full Range); unit: years] | 41.85 [23 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Maximum Tolerated Dose of Clofarabine When Administered in Combination With Alemtuzumab as Measured by CTC Version 3.0. (Phase 1)
Time Frame: 2 years
Population: Study enrolled six participants, but all participants withdrew or expired while on the study and study was ultimately terminated. As a results the study data was not collected and analyzed.
Arm/Group | Alemtuzumab and Clofarabine
Number analyzed (Participants) | 0

2. Primary Outcome: Number of Adverse Events
Time Frame: 2 years
Measure: Number; unit: adverse events
Arm/Group | Alemtuzumab and Clofarabine
Number analyzed (Participants) | 6
adverse events
  Nose Bleed | 1
  Diarrhea | 5
  Nausea | 6
  Vomiting | 6
  Dyspesia | 1
  Fever | 4
  Constipation | 5
  Pain | 6
  Insomnia | 6
  Itching | 4
  Anxiety | 6
  Rash | 1
  Hives | 1
  Dry Eyes | 1
  Deaths | 4

ADVERSE EVENTS:
Description: There is no longer access to participant level data for any Adverse Events collected in this study, therefore we report 0 participants at risk in this module. Please refer to Outcome Measure 2 where the available Adverse Event information for this study is reported
Arm/Group | Alemtuzumab and Clofarabine
All-Cause Mortality (participants affected / at risk) | 4/6
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Study enrolled six participants, but no participants completed study. Study was terminated due to slow accrual. All study data is reported by all participants since no data was analyzed due to study termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes